CLINICAL TRIAL: NCT04584645
Title: Increasing Influenza Vaccination in Individuals With Cardiovascular Conditions: Assessing the Effectiveness of a Digital Intervention in a Decentralized Randomized Controlled Trial
Brief Title: A Digital Flu Intervention for People With Cardiovascular Conditions
Acronym: CardioFlu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidation Health (Industry)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020/08/14
Record Dates: First submitted 2020-09-15; First posted 2020-10-14 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Diseases; Atrial Fibrillation; Abnormal Heart Rhythms; Cardiac Arrest; Heart Attack; Myocardial Infarction; Coronary Heart Disease; Heart Failure; Stroke; Cerebrovascular Accident
Keywords: Cardiovascular disease; Flu
MeSH Terms: conditions — Cardiovascular Diseases; Atrial Fibrillation; Arrhythmias, Cardiac; Heart Arrest; Myocardial Infarction; Coronary Disease; Heart Failure; Stroke; Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Masking Description: A set of existing Achievement members who have previously self-reported to meeting the inclusion criteria will be tagged for study inclusion, termed "participants". Since participants will be blinded to their study participation status, participants will not be asked to take any action to enroll in the study. In order to identify a target list of participants, Evidation Health will leverage already permissioned information from Achievement members, including data on their cardiovascular diagnoses, age, sex/gender, race/ethnicity, and country of residence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiovascular disorders digital intervention arm (CVD-I) (Experimental): Individuals with cardiovascular disease who receive a targeted digital intervention aimed at increasing influenza vaccination
  Interventions: Other: Targeted digital intervention
- cardiovascular disorders without digital intervention arm (No Intervention): Individuals with cardiovascular disease who receive no intervention

INTERVENTIONS:
Other: Targeted digital intervention — Messages that provide informational content on the influenza vaccine (sourced from the Centers for Disease Control and Prevention and the American Heart Association), specific information about influenza and cardiovascular disorders, and behavioral prompts (e.g., reminders) surrounding influenza vaccination behaviors.
  Arms: cardiovascular disorders digital intervention arm (CVD-I)

SUMMARY:
A 6-month prospective, digital randomized controlled trial targeting approximately 49,000 individuals to evaluate the effectiveness of an influenza vaccination intervention during influenza season for people with cardiovascular conditions

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Resides in the U.S.
* Speaks, reads, and understands English
* Has self-reported being diagnosed with any of the following cardiac conditions below in their Achievement profile:
* Atrial Fibrillation or Afib
* Abnormal or irregular heart rhythm, other arrhythmic heart disease
* Cardiac arrest, or heart attack (myocardial infarction)
* Coronary heart disease like a heart blockage, treated with medications, a stent in the heart, or sometimes bypass surgery-
* Heart failure, like congestive heart failure
* Stroke or cerebrovascular accident (CVA)

Exclusion Criteria:

* Participated in Step 1, Part 2 semi-structured interviews used to obtain feedback on the intervention messages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49138 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nell Marshall, DrPh, Principal Investigator — Evidation Health
Locations (1):
- Evidation Health, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dale LP, White L, Mitchell M, Faulkner G. Smartphone app uses loyalty point incentives and push notifications to encourage influenza vaccine uptake. Vaccine. 2019 Jul 26;37(32):4594-4600. doi: 10.1016/j.vaccine.2018.04.018. Epub 2018 Apr 23. PMID 29699784
- [Background] Dos Santos G, Tahrat H, Bekkat-Berkani R. Immunogenicity, safety, and effectiveness of seasonal influenza vaccination in patients with diabetes mellitus: A systematic review. Hum Vaccin Immunother. 2018;14(8):1853-1866. doi: 10.1080/21645515.2018.1446719. Epub 2018 Apr 9. PMID 29517396
- [Background] Doyle JD, Chung JR, Kim SS, Gaglani M, Raiyani C, Zimmerman RK, Nowalk MP, Jackson ML, Jackson LA, Monto AS, Martin ET, Belongia EA, McLean HQ, Foust A, Sessions W, Berman L, Garten RJ, Barnes JR, Wentworth DE, Fry AM, Patel MM, Flannery B. Interim Estimates of 2018-19 Seasonal Influenza Vaccine Effectiveness - United States, February 2019. MMWR Morb Mortal Wkly Rep. 2019 Feb 15;68(6):135-139. doi: 10.15585/mmwr.mm6806a2. PMID 30763298
- [Background] Frank L, Basch E, Selby JV; Patient-Centered Outcomes Research Institute. The PCORI perspective on patient-centered outcomes research. JAMA. 2014 Oct 15;312(15):1513-4. doi: 10.1001/jama.2014.11100. No abstract available. PMID 25167382
- [Background] Healthy People 2020. (2019). Retrieved from https://www.healthypeople.gov/. from Healthy People 2020, United States Department of Health and Human Services, Office of Disease Prevention and Health Promotion, https://www.healthypeople.gov/
- [Background] Hurley LP, Beaty B, Lockhart S, Gurfinkel D, Breslin K, Dickinson M, Whittington MD, Roth H, Kempe A. RCT of Centralized Vaccine Reminder/Recall for Adults. Am J Prev Med. 2018 Aug;55(2):231-239. doi: 10.1016/j.amepre.2018.04.022. Epub 2018 Jun 15. PMID 29910118
- [Background] Jackson ML, Chung JR, Jackson LA, Phillips CH, Benoit J, Monto AS, Martin ET, Belongia EA, McLean HQ, Gaglani M, Murthy K, Zimmerman R, Nowalk MP, Fry AM, Flannery B. Influenza Vaccine Effectiveness in the United States during the 2015-2016 Season. N Engl J Med. 2017 Aug 10;377(6):534-543. doi: 10.1056/NEJMoa1700153. PMID 28792867
- [Background] Lee WN, Stuck D, Konty K, Rivers C, Brown CR, Zbikowski SM, Foschini L. Large-scale influenza vaccination promotion on a mobile app platform: A randomized controlled trial. Vaccine. 2020 Apr 16;38(18):3508-3514. doi: 10.1016/j.vaccine.2019.11.053. Epub 2019 Nov 29. PMID 31787410
- [Background] Molinari NA, Ortega-Sanchez IR, Messonnier ML, Thompson WW, Wortley PM, Weintraub E, Bridges CB. The annual impact of seasonal influenza in the US: measuring disease burden and costs. Vaccine. 2007 Jun 28;25(27):5086-96. doi: 10.1016/j.vaccine.2007.03.046. Epub 2007 Apr 20. PMID 17544181
- [Background] Nehme EK, Delphia M, Cha EM, Thomas M, Lakey D. Promoting Influenza Vaccination Among an ACA Health Plan Subscriber Population: A Randomized Trial. Am J Health Promot. 2019 Jul;33(6):916-920. doi: 10.1177/0890117118823157. Epub 2019 Jan 10. PMID 30630342
- [Background] Rolfes MA, Flannery B, Chung JR, O'Halloran A, Garg S, Belongia EA, Gaglani M, Zimmerman RK, Jackson ML, Monto AS, Alden NB, Anderson E, Bennett NM, Billing L, Eckel S, Kirley PD, Lynfield R, Monroe ML, Spencer M, Spina N, Talbot HK, Thomas A, Torres SM, Yousey-Hindes K, Singleton JA, Patel M, Reed C, Fry AM; US Influenza Vaccine Effectiveness (Flu VE) Network, the Influenza Hospitalization Surveillance Network, and the Assessment Branch, Immunization Services Division, Centers for Disease Control and Prevention. Effects of Influenza Vaccination in the United States During the 2017-2018 Influenza Season. Clin Infect Dis. 2019 Nov 13;69(11):1845-1853. doi: 10.1093/cid/ciz075. PMID 30715278
- [Background] Samson, S., Lee, J., Tai, C., & Foschini, L. (2020, September). Digital intervention is effective at increasing influenza vaccination in people living with diabetes. Poster presented at the European Association for the Science of Diabetes in Vienna, Austria - Conference to occur digitally 22-25 September, 2020 due to COVID-19.
- [Background] Samson SI, Konty K, Lee WN, Quisel T, Foschini L, Kerr D, Liska J, Mills H, Hollingsworth R, Greenberg M, Beal AC. Quantifying the Impact of Influenza Among Persons With Type 2 Diabetes Mellitus: A New Approach to Determine Medical and Physical Activity Impact. J Diabetes Sci Technol. 2021 Jan;15(1):44-52. doi: 10.1177/1932296819883340. Epub 2019 Nov 20. PMID 31747789
- [Background] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Derived] Marshall NJ, Lee JL, Schroeder J, Lee WN, See J, Madjid M, Munagala MR, Piette JD, Tan L, Vardeny O, Greenberg M, Liska J, Mercer M, Samson S. Influence of Digital Intervention Messaging on Influenza Vaccination Rates Among Adults With Cardiovascular Disease in the United States: Decentralized Randomized Controlled Trial. J Med Internet Res. 2022 Oct 7;24(10):e38710. doi: 10.2196/38710. PMID 36206046
- See also: CDC Flu & Heart Disease and Stroke — https://www.cdc.gov/flu/highrisk/heartdisease.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A set of existing Achievement members who previously reported meeting the inclusion criteria were tagged for study inclusion. These participants were randomized using block randomization before being offered the opportunity to complete any study activities. Participants were sent offers via the Achievement platform to complete study activities. Participants could complete any number of survey activities. Completion of intervention activities was not required for enrollment for the CVD-I group.
Period: Overall Study
Arm/Group | Cardiovascular Disorders Digital Intervention Arm (CVD-I) | Cardiovascular Disorders Without Digital Intervention Arm
Started | 24570 | 24568
Completed | 5575 | 5662
Not Completed | 18995 | 18906
Not completed — Those participants who did not complete the 3 or 6 month surveys are considered "not completed". | 18995 | 18906

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiovascular Disorders Digital Intervention Arm (CVD-I) | Cardiovascular Disorders Without Digital Intervention Arm | Total
Number analyzed (Participants) | 5575 | 5662 | 11237
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (13.3) | 44.9 (13.5) | 44.95 (13.4)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participants had the option to select more than one response for Sex/Gender.
  Participants
    Woman | 4339 | 4427 | 8766
    Man | 1071 | 1114 | 2185
    Other | 169 | 135 | 304
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants had the option to select more than one response for Race/Ethnicity.
  Participants
    American Indian or Alaskan Native | 155 | 143 | 298
    Asian | 250 | 227 | 477
    Black or African American | 388 | 354 | 742
    Hispanic, Latino, or Spanish | 319 | 375 | 694
    Middle Eastern or North African | 46 | 50 | 96
    Native Hawaiian or Other Pacific Islander | 45 | 49 | 94
    White | 4510 | 4612 | 9122
    Another race or ethnicity not listed here | 60 | 64 | 124
    I prefer not to answer | 187 | 179 | 366
Has Health Insurance [Count of Participants; unit: Participants]
  Yes | 4815 | 4872 | 9687
  No | 343 | 368 | 711
  I don't know / I'm not sure | 50 | 53 | 103
  I prefer not to answer | 42 | 57 | 99
  No response | 325 | 312 | 637
Has a College Degree [Count of Participants; unit: Participants] | 3510 | 3381 | 6891
Household Income ≥ 75,000 [Count of Participants; unit: Participants] | 1909 | 1861 | 3770
Heart Conditions [Number; unit: participants] — Participants had the option to select more than one response for "Heart Conditions"
  participants
    Arrhythmia | 2251 | 2331 | 4582
    Atrial fibrillation | 488 | 496 | 984
    Cardiac arrest | 112 | 99 | 211
    Heart attack | 385 | 412 | 797
    Heart failure | 332 | 293 | 625
    Coronary heart disease | 366 | 356 | 722
    Stroke or CVA | 433 | 436 | 869
    Other cardiovascular diseases | 539 | 545 | 1084
    None of the above diagnoses | 1798 | 1844 | 3642

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Self-reported Influenza Vaccination Status as Vaccinated
Description: To determine the effectiveness of a digital intervention designed to increase influenza vaccination rates in individuals with cardiovascular diagnoses (CV diagnoses) by examining differences in self-reported influenza vaccination rates between individuals with cardiovascular disease who receive a targeted digital intervention (CVD-I) aimed at increasing influenza vaccination and those with CV diagnoses who received no intervention (CVD-C) by the end of the study period.
Time Frame: Up to 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiovascular Disorders Digital Intervention Arm (CVD-I) | Cardiovascular Disorders Without Digital Intervention Arm
Number analyzed (Participants) | 5575 | 5662
Participants | 3418 | 3355

2. Secondary Outcome: Number of Participants With Self-reported Influenza Vaccination Status as Vaccinated
Description: Differences in rates of self-reported influenza vaccination status after study start between individuals in the intervention group that completed different numbers of intervention messages (0 to 6 messages) over the course of the study
Time Frame: Up to 7 months
Population: This population consists of all individuals who are in the intervention arm and who have responded to the 3-month or 6-month survey.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Reported Influenza Vaccine After Completing 0 Interventions: Participants who Self-reported Influenza Vaccination After Study Start after interacting With 0 Intervention Messages Through Study Close
- Participants Who Reported Influenza Vaccine After Completing 1 Intervention: Participants who Self-reported Influenza Vaccination After Study Start after interacting With 1 Intervention Message Through Study Close
- Participants Who Reported Influenza Vaccine After Completing 2 Interventions: Participants who Self-reported Influenza Vaccination After Study Start after interacting With 2 Intervention Messages Through Study Close
- Participants Who Reported Influenza Vaccine After Completing 3 Interventions: Participants who Self-reported Influenza Vaccination After Study Start after interacting With 3 Intervention Messages Through Study Close
- Participants Who Reported Influenza Vaccine After Completing 4 Interventions: Participants who Self-reported Influenza Vaccination After Study Start after interacting With 4 Intervention Messages Through Study Close
- Participants Who Reported Influenza Vaccine After Completing 5 Interventions: Participants who Self-reported Influenza Vaccination After Study Start after interacting With 5 Intervention Messages Through Study Close
- Participants Who Reported Influenza Vaccine After Completing 6 Interventions: Participants who Self-reported Influenza Vaccination After Study Start after interacting With 6 Intervention Messages Through Study Close
Arm/Group | Participants Who Reported Influenza Vaccine After Completing 0 Interventions | Participants Who Reported Influenza Vaccine After Completing 1 Intervention | Participants Who Reported Influenza Vaccine After Completing 2 Interventions | Participants Who Reported Influenza Vaccine After Completing 3 Interventions | Participants Who Reported Influenza Vaccine After Completing 4 Interventions | Participants Who Reported Influenza Vaccine After Completing 5 Interventions | Participants Who Reported Influenza Vaccine After Completing 6 Interventions
Number analyzed (Participants) | 424 | 354 | 392 | 455 | 592 | 837 | 2476
Participants | 211 | 184 | 245 | 276 | 355 | 510 | 1612

3. Secondary Outcome: Participant Completion Rate
Description: Differences in completion rates of specific intervention types by individuals in the group receiving the targeted intervention
Time Frame: Up to 7 months
Population: Participants in the intervention arm who received and responded to either the 3 or 6 month survey.
Measure: Count of Participants; unit: Participants
Groups:
- Completion Rate of Educational Videos: Percentage of Participants that Completed the Intervention "Educational Videos"
- Completion Rate of Knowledge Quiz: Percentage of Participants that Completed the Intervention "Knowledge Quiz"
- Completion Rate of Cost Article: Percentage of Participants that Completed the Intervention "Cost Article"
- Completion Rate of CDC Heart-Focused Article: Percentage of Participants that Completed the Intervention "CDC Heart-Focused Article"
- Completion Rate of Location Finder: Percentage of Participants that Completed the Intervention "Location Finder"
- Completion Rate of Date Setter: Percentage of Participants that Completed the Intervention "Date Setter"
Arm/Group | Completion Rate of Educational Videos | Completion Rate of Knowledge Quiz | Completion Rate of Cost Article | Completion Rate of CDC Heart-Focused Article | Completion Rate of Location Finder | Completion Rate of Date Setter
Number analyzed (Participants) | 5531 | 5531 | 5531 | 5531 | 5531 | 5531
Participants | 3789 | 4216 | 4243 | 4283 | 3740 | 3682

4. Secondary Outcome: Self-Reported Influenza Vaccination Status Prediction
Description: Development of a logistic regression model to predict self-reported influenza vaccination status using vaccination predictors such as vaccine drivers/barriers, and vaccine knowledge.
Time Frame: Up to 7 months
Measure: Mean (95% Confidence Interval); unit: Odds ratio of influenza vaccination
Groups:
- Influenza Vaccine Offered: The health behavior "Influenza Vaccine Offered" as a predictor of influenza vaccination
- High Risk Group Informed: The health behavior "High Risk Group Informed" as a predictor of influenza vaccination
- Sees Primary Care Physician: The health behavior "Sees Primary Care Physician" as a predictor of influenza vaccination
- Hospitalized: The health behavior "Hospitalized" as a predictor of influenza vaccination
- Sees Cardiologist: The health behavior "Sees Cardiologist" as a predictor of influenza vaccination
Arm/Group | Influenza Vaccine Offered | High Risk Group Informed | Sees Primary Care Physician | Hospitalized | Sees Cardiologist
Number analyzed (Participants) | 11237 | 11237 | 11237 | 11237 | 11237
Odds ratio of influenza vaccination | 11.2 [10.14 to 12.36] | 2.37 [2.17 to 2.59] | 1.9 [1.76 to 2.06] | 1.89 [1.57 to 2.27] | 1.63 [1.48 to 1.81]

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: Adverse Events were not collected or assessed as part of this study.
Arm/Group | Cardiovascular Disorders Digital Intervention Arm (CVD-I) | Cardiovascular Disorders Without Digital Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT04584645/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04584645/SAP_000.pdf